CLINICAL TRIAL: NCT04595448
Title: Lymphatic Function in Patients With Secondary Tricuspid Valve Regurgitation - An Unknown Collaborator in a System Under Pressure
Brief Title: Lymphatic Function in Patients With Secondary Tricuspid Valve Regurgitation
Acronym: LYMTRIVA
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-113-20
Record Dates: First submitted 2020-09-18; First posted 2020-10-20 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2022-05

CONDITIONS: Lymphatic Insufficiency; Heart Failure; Edema
MeSH Terms: conditions — Heart Failure; Edema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients suffering from moderate tricuspid valve regurgitation
- Controls: Cardiovascular healthy, age, gender and weight matched controls.

SUMMARY:
The study will examine the lymphatic functional and morphological status in patients with moderate tricuspid valve regurgitation compared to healthy age and gender-matched controls.

The study will use t2 weighted MRI, Near-infrared fluorescence imaging, and plethysmography to examine the above-mentioned question.

DETAILED DESCRIPTION:
The study will examine the lymphatic functional and morphological status in patients with moderate tricuspid valve regurgitation compared to healthy age and gender-matched controls.

Subjects will be examined at one occasion using t2-weighted MRIs to evaluated lymphatic anatomy and Near-infrared fluorescence imaging for evaluation of superficial peripheral lymphatic function. Finally, the capillary filtration rate will be estimated using plethysmography.

ELIGIBILITY:
Patients:

Inclusion criteria:

* Patients with moderate to severe tricuspid regurgitation
* Age ≥18 years
* Informed consent

Exclusion criteria:

* Reduced ejection fraction (<50%)
* Congenital heart disease
* Left sided valve disease
* MRI contraindications (All metal implants, cochlear implants, pacemakers etc.)
* Claustrophobia
* Peripheral edema
* BMI>30
* Age<18.

Controls:

Inclusion criteria:

* Healthy
* Age ≥18 years
* Age, gender and weight matched with included patients.

Exclusion criteria:

* Cardiovascular disease
* MRI contraindications (All metal implants, cochlear implants, pacemakers etc.)
* Claustrophobia
* Peripheral edema
* BMI>30
* Age<18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe tricuspid regurgitation and healthy, age, gender, and weight-matched controls
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Thoracic duct tortuosity (centimeters/centimeters) | 20 minutes
  Based on MRI, the thoracic duct will be rendered and measured with regards to tortuosity (full length/straight length)
Thoracic duct volume (cubic centimetres) | 30 minutes
  Based on MRI, the thoracic duct will be rendered and measured with regards to volume.
Excess fluid (yes/no) | 40 minutes
  Based on MRI, the existence of excess fluid in the pericardial, thoracic and abdominal cavity will be accessed.
Peripheral lymphatic velocity (centimeters/second) | 1 hour
  Peripheral lymphatic fluid velocity (centimeters/second) will be calculated based upon NIRF sequences.
Peripheral lymphatic frequency (contractions/minute) | 1 hour 30 minutes
  Peripheral lymphatic contraction frequency (contractions/minute) will be calculated based upon NIRF sequences.

SECONDARY OUTCOMES:
Capillary filtration | 2 hours
  Evaluation of capillary filtration rate estimated using plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Aarhus N, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No